CLINICAL TRIAL: NCT00530413
Title: Study of Phenobarbital Inhibition of Catamenial Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB needs updated
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xUTHSC-07
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Phenobarbital - dose based by weight range
  Interventions: Drug: Phenobarbital
- 2 (Placebo Comparator): Placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phenobarbital — Phenobarbital will be given based on weight range
  Arms: 1
Other: Placebo — Placebo group
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness of low-dose Phenobarbital on the treatment of catamenial epilepsy.

We propose that since the catamenial seizures are associated with the reduction in levels of GABA-enhancing allopregnanolone, short-term replacement with the GABAR-enhancing agent Phenobarbital will reduce the incidence of catamenial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients seeking medical attention for seizures
* Regular menstrual cycles
* At least 2 seizures per month
* Must be on at least one form of birth control other than abstinence
* Must be on a stable anticonvulsant regimen of at least one and not exceeding three anticonvulsants, and not be using any perimenstrual seizure medications of hormone preparations
* If taking benzodiazepines for therapeutic purposes, must be on a stable regular dose
* Must be willing to take at least 400mcg of folic acid a day while in the study
* Must be able to detect, count or record seizures

Exclusion Criteria:

* Can not be pregnant or trying to become pregnant
* Can not have used hormonal birth control methods for at least 3 months prior to enrollment
* Can not have an allergy to Phenobarbital
* Can not have a history of non-epileptic seizures
* Can not have a know liver dysfunction or history of chronic hepatitis
* Can not have a history of neurological disorder or history of status epilepticus in the preceding year
* Can not ahve a physical or psychiatric condition which in the PIs opinion could compromise her ability to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Screening, 3 month and final visit
Depression Epworth Sleepiness Scale (ESS) | Screening, 3 month and final visit
Quality of Life in Epilepsy (QOLIE-10) | Screening, 3 month and Final Visit
Addenbrooke's Cognitive Examination (ACE) | Screening, 3 month and Final Visit

SECONDARY OUTCOMES:
Determine tolerance of medication using the depression, cognitive and sleepiness screening tools listed above | Screening, 3 months, final visit

CONTACTS AND LOCATIONS:
Overall Officials: Lazar J Greenfield, Jr, MD, PhD, Principal Investigator — University of Toledo Health Science Campus
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States